CLINICAL TRIAL: NCT00274612
Title: A Prospective Randomised Open- Label Blinded-Endpoint (PROBE) Trial Comparing Telmisartan (MICARDIS®) (40-80-80mg QD) and Ramipril (2.5-5--10mg QD) in Patients With Mild-to-Moderate Hypertension Using Ambulatory Blood Pressure Monitoring. PRISMA = Prospective Randomised Investigation of the Safety and Efficacy of Micardis® vs Ramipril Using ABPM
Brief Title: Prospective Randomised Investigation of the Safety and Efficacy of Micardis® vs Ramipril Using ABPM
Acronym: PRISMA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 502.391
Record Dates: First submitted 2006-01-10; First posted 2006-01-11 (Estimated); Last update posted 2013-11-01 (Estimated); Status verified 2013-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Telmisartan; Ramipril

INTERVENTIONS:
Drug: Telmisartan
Drug: Ramipril

SUMMARY:
The primary objective of this study is to demonstrate that telmisartan 80 mg (MICARDIS®) is at least as effective and possibly superior to ramipril 5mg and 10mg in lowering mean ambulatory diastolic blood pressure (DBP) and systolic blood pressure (SBP) during the last 6 hours of the 24-hour dosing interval in mild-to-moderate hypertensive patients at the end of an 8 and 14-week treatment period, respectively.

DETAILED DESCRIPTION:
Secondary objectives will compare telmisartan (80 mg) (MICARDIS® and ramipril (5 mg and 10 mg) on: 1) the reduction in the last 6-hour ABPM mean pulse pressure (PP) relative to dosing, 2) the reductions in the 24-hour ABPM mean DBP, SBP and PP relative to dosing, 3) reductions in ABPM mean DBP, SBP and PP during other periods of the 24-hour dosing interval (i.e., morning, daytime, and nighttime) relative to clock time, 4) change from baseline in systolic and diastolic blood pressure load during the 24-hour dosing interval, 5) reductions in the mean seated trough DBP and SBP measured using a manual in-clinic cuff sphygmomanometer, 6) responder rates as determined by both ABPM and manual in-clinic cuff measurements and 7) Health-Related Quality of Life (HRQL).

Study Hypothesis:

It is hypothesised that the rise of blood pressure (BP) during the last hours of the sleeping period is a cause of the high incidence of cardiovascular events in the morning. The purpose of the present study is to demonstrate that telmisartan (MICARDIS®) is not inferior to ramipril in lowering blood pressure in patients with mild-to-moderate hypertension. Blood pressure will be assessed by ambulatory blood pressure monitoring (ABPM) as this will allow comparison of the full 24-hour effects of both treatments without artefacts (e.g., white-coat hypertension) introduced by measurement of blood pressure in the clinic. This will measure diastolic blood pressures over the entire 24-hour dosing interval, with primary attention focused on the last six hours of the dosing interval.

NULL AND ALTERNATIVE HYPOTHESES In order to test the multiple hypotheses (e.g., non-inferiority and superiority of telmisartan compared to ramipril), multiple dosages (i.e., telmisartan 80mg (MICARDIS®) versus ramipril 5mg and ramipril 10mg after 8 and 14 weeks of treatment, respectively), and the two endpoints (i.e., reduction in DBP and SBP during the last 6 hours of the 24-hour dosing interval) as measured by ABPM, a completely hierarchical, closed testing procedure will be used.

Hierarchical Closed Testing Procedure:

1. Non-inferiority of telmisartan 80 mg (MICARDIS®) compared to ramipril 5 mg at the end of the 8 week treatment period in the reduction of DBP during the last 6 hours of the 24 hour dosing interval; if significant then,
2. Superiority of telmisartan 80 mg (MICARDIS®) compared to ramipril 5 mg at the end of the 8-week treatment period in the reduction of DBP during the last 6 hours of the 24-hour dosing interval; if significant then,
3. Superiority of telmisartan 80mg (MICARDIS®) compared to ramipril 5 mg at the end of the 8-week treatment period in the reduction of SBP during the last 6 hours of the 24-hour dosing interval; if significant then,
4. Non-inferiority of telmisartan 80mg (MICARDIS®) compared to ramipril 10 mg at the end of an 14 week treatment period in the reduction of DBP during the last 6 hours of the 24-hour dosing interval; if significant then,
5. Superiority of telmisartan 80mg (MICARDIS®) compared to ramipril 10 mg at the end of an 14-week treatment period in the reduction of DBP during the last 6 hours of the 24-hour dosing interval; and if significant then,
6. Superiority of telmisartan 80mg (MICARDIS®) compared to ramipril 10mg at the end of an 14-week treatment period in the reduction of SBP during the last 6 hours of the 24-hour dosing interval.

A difference of 2 mmHg was determined to be the maximum difference between the mean reductions in DBP during the last 6 hours of the 24-hour dosing interval for the two treatments which would be considered to have no clinical importance (i.e., the limit for non inferiority). Thus non-inferiority of telmisartan compared to ramipril will be tested using the following set of hypotheses:

Null Hypothesis:

The overall mean reduction from baseline in ABPM mean DBP during the last 6 hours of the 24-hour dosing interval for telmisartan 80 mg (MICARDIS®) is inferior to that for ramipril by at least 2 mmHg.

Alternative Hypothesis: The overall mean reduction from baseline in ABPM mean DBP during the last 6 hours of the 24-hour dosing interval for telmisartan 80mg (MICARDIS®) is less than 2 mmHg smaller than that for ramipril.

These hypotheses can be stated as:

H0: dT - dR less than or equal to -2 mmHg versus HA: dT - dR > -2 mmHg where dT and dR represent the overall mean reduction from baseline in ABPM mean DBP during the last 6 hours of the 24-hour dosing interval for telmisartan and ramipril, respectively, adjusted for any other factors included in the statistical model.

If the lower limit of the two-sided 95% confidence interval for the difference between the least square means of both treatments (telmisartan - ramipril) lies above -2 mmHg, then it will be concluded that telmisartan 80mg (MICARDIS®) is at least as effective as ramipril (5mg after 8 weeks of treatment or 10mg after 14 weeks of treatment, depending upon the comparison) in reducing DBP during the last 6 hours of the 24-hour dosing interval.

Superiority of telmisartan (MICARDIS®) compared to ramipril will be tested using the following set of hypotheses:

Null Hypothesis:

The overall mean reduction from baseline in the ABPM mean during the last 6 hours of the 24-hour dosing interval for telmisartan 80mg (MICARDIS®) is less than or equal to that for ramipril.

Alternative Hypothesis: The overall mean reduction from baseline in the ABPM mean during the last 6 hours of the 24-hour dosing interval for telmisartan 80mg (MICARDIS®) is greater than that for ramipril.

These hypotheses can be stated as:

H0: dT - dR less than or equal to 0 mmHg versus HA: dT - dR > 0 mmHg where dT and dR represent the overall mean reduction from baseline in ABPM mean DBP during the last 6 hours of the 24-hour dosing interval for telmisartan and ramipril, respectively, adjusted for any other factors included in the statistical model.

If the lower limit of the two-sided 95% confidence interval for the difference between the least square means of both treatments (telmisartan (MICARDIS®) - ramipril) is greater than zero, then it will be concluded that telmisartan 80mg (MICARDIS®) is statistically superior to ramipril (5mg after 8 weeks of treatment or 10mg after 14 weeks of treatment, depending upon the comparison) in reducing blood pressure (DBP or SBP, depending upon the comparison) during the last 6 hours of the 24-hour dosing interval.

Comparison(s):

Reductions in blood pressure during the last 6 hours of the 24-hour dosing interval as measured by ABPM in patients treated with telmisartan (MICARDIS®) compared to patients treated with ramipril. The primary analysis will consist of a closed testing procedure first testing for non-inferiority of telmisartan 80mg (MICARDIS®) compared to ramipril 10mg after fourteen weeks of treatment in the reduction in diastolic blood pressure (DBP); if significant, testing for superiority of telmisartan 80 mg (MICARDIS®) compared to ramipril 10 mg in the reduction in DBP; if significant, testing for superiority of telmisartan 80 mg (MICARDIS®) compared to ramipril 10 mg in the reduction of systolic blood pressure (SBP); if significant, testing for non-inferiority of telmisartan 80 mg (MICARDIS®) compared to ramipril 5 mg after eight weeks of treatment in the reduction in DBP; if significant, testing for superiority of telmisartan 80 mg (MICARDIS®) compared to ramipril 5 mg in the reduction in DBP; and if significant, testing for superiority of telmisartan 80mg (MICARDIS®) compared to ramipril 5mg in the reduction in SBP.

ELIGIBILITY:
Inclusion Criteria:

1. Mild-to-moderate hypertension defined as a mean seated diastolic blood pressure of greater than or equal to 95 mmHg and less than or equal to 109 mmHg, measured by manual cuff sphygmomanometer at Visit 2.
2. 24-hour mean DBP of greater than or equal to 85 mmHg at Visit 3 as measured by ABPM.
3. Age 18 years or older.
4. Ability to stop any current antihypertensive therapy without risk to the patient (investigator's discretion).
5. Ability to provide written informed consent in accordance with GCP and local legislation.

Exclusion Criteria:

1. Pre-menopausal women (last menstruation approximately less than or equal to 1 year prior to signing informed consent) who:

   * Are not surgically sterile
   * Are nursing,
   * Are of child-bearing potential and are NOT practicing acceptable methods of birth control, or do NOT plan to continue practicing an acceptable method throughout the study. Acceptable methods of birth control include intra uterine device, oral, implantable or injectable contraceptives.
2. Night shift workers who routinely sleep during the daytime and whose work hours include midnight to 4:00 A.M.
3. Mean sitting SBP greater than or equal to180 mmHg or mean sitting DBP greater than or equal to 110 mmHg during any visit of the placebo run-in period.
4. Known or suspected secondary hypertension (i.e., pheochromocytoma).
5. Hepatic and/or renal dysfunction as defined by the following laboratory parameters:

   * SGPT (ALT) or SGOT (AST) > 2 times the upper limit of normal range.
   * Serum creatinine > 2.3mg/dL (or > 203 micromol/l).
6. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney.
7. Clinically relevant sodium depletion, hypokalaemia or hyperkalaemia.
8. Uncorrected volume depletion.
9. Primary aldosteronism.
10. Hereditary fructose intolerance.
11. Biliary obstructive disorders.
12. Congestive heart failure (NYHA functional class CHF III-IV).
13. Unstable angina within the past three months prior to start of run in period.
14. Stroke within the past six months prior to start of run in period.
15. Myocardial infarction or cardiac surgery within the past three months prior to start of run in period.
16. PTCA (percutaneous transluminal coronary angioplasty) within the past three months prior to start of run in period.
17. Sustained ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the investigator.
18. Hypertrophic obstructive cardiomyopathy, aortic stenosis, haemodynamically relevant stenosis of the aortic or mitral valve.
19. Patients with insulin-dependent diabetes mellitus whose diabetes has not been stable and controlled for at least the past three months as defined by an HbA1C greater than or equal to 10%.
20. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin II receptor antagonists.
21. History of drug or alcohol dependency within 6 months prior to start of run in period.
22. Concomitant administration of any medications known to affect blood pressure, except medication allowed by the protocol.
23. Any investigational therapy within one month of start of run in period.
24. Known hypersensitivity to any component of the formulations.
25. Any clinical condition which, in the opinion of the investigator would not allow safe completion of the protocol and safe administration of trial medication.
26. Inability to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 801
Dates: Start 2002-10; Primary Completion 2003-11 (Actual); Study Completion 2003-11

PRIMARY OUTCOMES:
Changes in the last 6-hour mean (relative to dose time) diastolic and systolic blood pressure (DBP and SBP) as measured by ABPM | after 8 and 14 weeks

SECONDARY OUTCOMES:
Changes in the last 6-hour ABPM mean (relative to dosing time) for pulse pressure (PP) | after 8 and 14 weeks
Changes in the 24-hour ABPM mean (relative to dosing time) for DBP, SBP and PP | after 8 and 14 weeks
Changes in the ABPM mean (relative to clock-time) for DBP, SBP and PP during the morning, daytime and night-time periods of the 24-hour dosing interval. | after 8 and 14 weeks
Changes in SBP and DBP load during the 24-hour dosing interval | after 8 and 14 weeks
Changes in mean seated trough DBP and SBP as measured by manual in-clinic cuff sphygmomanometer | after 8 and 14 weeks
Responder rates based on both the 24-hour ABPM mean (relative to dose time) BPs and manual in-clinic trough cuff measurements | after 8 and 14 weeks
Changes from baseline in patient Health Related Quality of Life (HRQL) as measured by Psychological General Wellbeing Index (PGWB). | week 8 and 14
Manually triggered BP measurements before going to bed and upon arising in the morning | after 8 and 14 weeks
Incidence of adverse events | up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim Ltd./Bracknell
Locations (60):
- Austria (6):
  - Rehabilitationszentrum für Herz- und Kreislauferkrankungen, Bad Tatzmannsdorf
  - A.ö. Landeskrankenhaus Bruck a. d. Mur, Bruck A. D. Mur
  - Landeskrankenhaus Graz West, Graz
  - Medizinische Universitätsklinik Graz, Graz
  - Univ.-Klinik für Innere Medizin III, Vienna
  - Landeskrankenhaus Villach, Villach
- France (6):
  - Boehringer Ingelheim Investigational Site, Angers
  - Hôpital Saint André, Bordeaux
  - Boehringer Ingelheim Investigational Site, Laval
  - Boehringer Ingelheim Investigational Site, Mayenne
  - Boehringer Ingelheim Investigational Site, Saint Laurent Du Medoc
  - Boehringer Ingelheim Investigational Site, Saumur
- Germany (9):
  - Boehringer Ingelheim Investigational Site, Gaggenau
  - Boehringer Ingelheim Investigational Site, Haag
  - Boehringer Ingelheim Investigational Site, Linkenheim-Hochstetten
  - Boehringer Ingelheim Investigational Site, Mühldorf
  - Boehringer Ingelheim Investigational Site, Plattling
  - Boehringer Ingelheim Investigational Site, Unterschneidheim
  - Boehringer Ingelheim Investigational Site, Villingen-Schwenningen
  - Boehringer Ingelheim Investigational Site, Vilsbiburg
  - Boehringer Ingelheim Investigational Site, Westerkappeln
- Netherlands (4):
  - Boehringer Ingelheim Investigational Site, Bennebroek
  - Boehringer Ingelheim Investigational Site, Heerlen
  - Boehringer Ingelheim Investigational Site, Nijverdal
  - Boehringer Ingelheim Investigational Site, Rotterdam
- South Africa (4):
  - Boehringer Ingelheim Investigational Site, Bellville
  - Health Emporium, Midrand
  - Boehringer Ingelheim Investigational Site, Vanderbijlpark
  - 1 Military Hospital, Vootrekkehoogte
- Spain (7):
  - Boehringer Ingelheim Investigational Site, Barcelona
  - Hospital de Galdakao, Galdakao / Vizcaya
  - Pabellon de Consultas, Madrid
  - Edificio de Consultas Externas, Oviedo
  - Boehringer Ingelheim Investigational Site, Salamanca
  - Pabellon B / 1 piso, Santa Coloma de Gramanet
  - Centro de Diagnostico y Tratamiento, Seville
- Switzerland (6):
  - Universitätsspital Basel, Basel
  - Boehringer Ingelheim Investigational Site, Basel
  - Schweizerisches Herz- und Gefässzentrum, Bern
  - Cardiocentro Ticino, Lugano
  - Boehringer Ingelheim Investigational Site, Muralto
  - Boehringer Ingelheim Investigational Site, Münsterlingen
- United Kingdom (18):
  - Boehringer Ingelheim Investigational Site, Ashford
  - Boehringer Ingelheim Investigational Site, Atherstone
  - Boehringer Ingelheim Investigational Site, Bath
  - Boehringer Ingelheim Investigational Site, Bedworth
  - Boehringer Ingelheim Investigational Site, Coventry
  - Boehringer Ingelheim Investigational Site, Doncaster
  - Boehringer Ingelheim Investigational Site, Fowey
  - Boehringer Ingelheim Investigational Site, Frome
  - Boehringer Ingelheim Investigational Site, Glasgow
  - Boehringer Ingelheim Investigational Site, Ilford
  - Boehringer Ingelheim Investigational Site, Lesley
  - Boehringer Ingelheim Investigational Site, Lostwithiel
  - Boehringer Ingelheim Investigational Site, Royal Leamington Spa
  - Boehringer Ingelheim Investigational Site, Ryde
  - Boehringer Ingelheim Investigational Site, Trowbridge
  - Boehringer Ingelheim Investigational Site, Wells Next to the Sea
  - Boehringer Ingelheim Investigational Site, Whitstable
  - York District Hospital, York